CLINICAL TRIAL: NCT04696887
Title: TechSAge Tele Tai Chi for People Aging With Mobility Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: University of Illinois at Urbana-Champaign (Other); University of Georgia (Other); Tai Chi for Health Institute (Unknown); National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Principal Investigator, Tracy Mitzner, Senior Research Scientist, Georgia Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H19560
Record Dates: First submitted 2020-12-15; First posted 2021-01-06 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Aging; Disability Physical
Keywords: mind-body exercise; tai chi; technology

STUDY DESIGN:
Intervention Model Description: All participants will be screened and assigned to the same condition in a phased/rolling enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tele Tai Chi (Experimental): 8-week Tele Tai Chi intervention
  Interventions: Behavioral: Tele Tai Chi Intervention for Persons Aging with Long-Term Mobility Disabilities

INTERVENTIONS:
Behavioral: Tele Tai Chi Intervention for Persons Aging with Long-Term Mobility Disabilities — • 8-week Tele Tai Chi intervention, participants will use a tablet or computer to join a small-group, online class (1hr, twice weekly) from home; during each session, participants will exercise as a group along with the pre-recorded video lessons and have the opportunity for social interaction (via video chat) before and after class.
  Other Names: Seated Tai Chi for Arthritis

SUMMARY:
This study uses videoconferencing to deliver an evidence-based exercise program, Seated Tai Chi for Arthritis, to adults aging with long-term mobility disabilities. In the 8-week Tele Tai Chi intervention, participants will use a tablet or computer to join a small-group, online class (1hr, twice weekly) from home; during each session, participants will exercise as a group along with the pre-recorded video lessons and have the opportunity for social interaction (via video chat) before and after class. The study will examine the effects of the Tele Tai Chi program on physical activity and social connectedness for adults aging with long-term mobility disabilities, a population likely to experience barriers to exercise participation.

DETAILED DESCRIPTION:
This study is part of the Rehabilitation Engineering Research Center on Technologies to Support Aging-in-Place for People with Long-Term Disabilities (RERC TechSAge). This study uses videoconferencing to translate an evidence-based exercise program for older adults, Seated Tai Chi for Arthritis, from an in-person setting to a remote class and to a different population, adults aging with mobility disabilities. In the 8-week Tele Tai Chi intervention, participants will use a tablet or computer to join a small-group, online class (1hr, twice weekly) from home; during each session, participants will exercise as a group along with the pre-recorded video lessons and have the opportunity for social interaction (via video chat) before and after class. The study will examine the effects of the Tele Tai Chi program on physical activity and social connectedness (primary outcomes), as well as exercise self-efficacy, falls efficacy, depression, quality of life, and pain (secondary outcomes) for adults aging with long-term mobility disabilities, a population likely to experience barriers to in-person exercise participation.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 60-80
* Self-identify as having a mobility disability, use a mobility aid (i.e., cane, crutches, wheelchair, walker, or scooter) or have serious difficulty walking or climbing stairs
* Mobility disability for at least 10 years
* Passing score on Physical Activity Readiness Questionnaire (PAR-Q) or letter from physician stating approved to participate in the intervention
* Passing score on Telephone Interview for Cognitive Status (TICS)-score 26 and above included
* Passing score of brief Technology Proficiency Screen (e.g., be able to do send and receive email)
* Have access to a webcam on computer or tablet
* Plan to have internet access for six months from screening
* Live in the US
* Be conversational in English
* Available to attend 1 hr online class 2x a week for 8 weeks

Exclusion Criteria:

* Blind or deaf
* Significant Tai Chi practice during the past 6 months

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Physical activity | Baseline, Week 1-8 of intervention, Post-Intervention (8 week assessment), 1 month follow-up
  Change in physical activity (mode, frequency, duration, intensity) as measured by the leisure activity dimension of the Physical Activity Scale for Persons with Physical Disabilities1, a self-report measure of physical activity (Range 0-98.67; Higher score means greater physical activity. Lower score means less physical activity). Self-report completion of Tai Chi practice (Range 1-4; Higher score indicates greater frequency of practice. Lower score indicates less frequent of practice).
Social connectedness | Baseline, Post-Intervention (8 week assessment), 1 month follow-up
  Change in perception of social connectedness (loneliness), as measured by the UCLA Loneliness Scale (ULS-8)3 (Range 8-32; Higher score indicates a greater degree of loneliness. Lower score reflects a lower degree of loneliness), Social Isolation Questionnaire4 (Social Disconnectedness Scale, Social Isolation Scale, Perceived Social Isolation scale; Range 15-67; Higher score indicates a greater degree of loneliness. Lower score reflects a lower degree of loneliness).

SECONDARY OUTCOMES:
Exercise Self-Efficacy | Baseline, Post-Intervention (8 week assessment), 1 month follow-up
  Change in confidence in being able to exercise, as measured by the Exercise Self-Efficacy Scale (ESES) Scale5. A higher score indicates a greater confidence in being able to exercise. A lower score reflects less confidence in being able to exercise. Range (10-40).
Falls Efficacy | Baseline, Post-Intervention (8 week assessment), 1 month follow-up
  Change in confidence in being able to engage in activities without falling, as measured by the Falls Efficacy Scale6 (Range 10-100; Lower score indicates greater confidence in being able to engage in activities without falling. Higher score reflects less confidence in being able to engage in activities without falling; Total score of greater than 70 indicates that the person has a fear of falling), and a 3-item indicator of fear of falling (adapted from7-8; Range 0-5; Lower score indicates less fear of falling. Higher score reflects greater fear of falling).
Depression | Baseline, Post-Intervention (8 week assessment), 1 month follow-up
  Change in emotional distress (depression), as measured by the PROMIS Emotional Distress - Depression - Short Form9. Higher score means greater emotional distress. A lower score means less emotional distress. Range (8-40).
Quality of Life (QOL) | Baseline, Post-Intervention (8 week assessment), 1 month follow-up
  Change in self-reported quality of life, as measured by the Kemp Quality of Life single item scale10. Higher score means higher quality of life. A lower score means lower quality of life. Range (1-7).
Pain Interference | Baseline, PPost-Intervention (8 week assessment), 1 month follow-up
  Change in pain interference, as measured the PROMIS Pain Interference - Short Form11. Higher score means greater pain interference. A lower score means less pain interference. Range (4-20).

OTHER OUTCOMES:
Technology Acceptance | Baseline, Post-Intervention (8 week assessment)
  Change in technology acceptance, as measured the Technology Acceptance Questionnaire (modified12,13,14). Higher score means greater technology acceptance. A lower score means less greater technology acceptance. Range (20-140).
Physical Activity Class Satisfaction | Post-Intervention (8 week assessment)
  Class Satisfaction as measured by the dimensions of mastery experience, teaching, interaction with others, improvement of health and fitness, and relaxation from the Physical Activity Class Satisfaction Questionnaire2, a self-report measure of satisfaction related to exercise classes (Range 22-176); Higher score means greater satisfaction with physical activity class.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Inclusive Design and Innovation, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Washburn RA, Zhu W, McAuley E, Frogley M, Figoni SF. The physical activity scale for individuals with physical disabilities: development and evaluation. Arch Phys Med Rehabil. 2002 Feb;83(2):193-200. doi: 10.1053/apmr.2002.27467. PMID 11833022
- [Result] 2Cunningham, G. B. (2020). Development of the Physical Activity Class Satisfaction Questionnaire (PACSQ). Measurement in Physical Education and Exercise Science, 11(3), 161-176.
- [Result] Hays RD, DiMatteo MR. A short-form measure of loneliness. J Pers Assess. 1987 Spring;51(1):69-81. doi: 10.1207/s15327752jpa5101_6. PMID 3572711
- [Result] Cornwell EY, Waite LJ. Measuring social isolation among older adults using multiple indicators from the NSHAP study. J Gerontol B Psychol Sci Soc Sci. 2009 Nov;64 Suppl 1(Suppl 1):i38-46. doi: 10.1093/geronb/gbp037. Epub 2009 Jun 9. PMID 19508982
- [Result] Kroll T, Kehn M, Ho PS, Groah S. The SCI Exercise Self-Efficacy Scale (ESES): development and psychometric properties. Int J Behav Nutr Phys Act. 2007 Aug 30;4:34. doi: 10.1186/1479-5868-4-34. PMID 17760999
- [Result] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Result] Finlayson M, Peterson EW, Cho C. Pilot study of a fall risk management program for middle aged and older adults with MS. NeuroRehabilitation. 2009;25(2):107-15. doi: 10.3233/NRE-2009-0505. PMID 19822941
- [Result] Walker JE, Howland J. Falls and fear of falling among elderly persons living in the community: occupational therapy interventions. Am J Occup Ther. 1991 Feb;45(2):119-22. doi: 10.5014/ajot.45.2.119. PMID 2035588
- [Result] Pilkonis PA, Choi SW, Reise SP, Stover AM, Riley WT, Cella D; PROMIS Cooperative Group. Item banks for measuring emotional distress from the Patient-Reported Outcomes Measurement Information System (PROMIS(R)): depression, anxiety, and anger. Assessment. 2011 Sep;18(3):263-83. doi: 10.1177/1073191111411667. Epub 2011 Jun 21. PMID 21697139
- [Result] Siebens HC, Tsukerman D, Adkins RH, Kahan J, Kemp B. Correlates of a Single-Item Quality-of-Life Measure in People Aging with Disabilities. Am J Phys Med Rehabil. 2015 Dec;94(12):1065-74. doi: 10.1097/PHM.0000000000000298. PMID 25888654
- [Result] Amtmann D, Cook KF, Jensen MP, Chen WH, Choi S, Revicki D, Cella D, Rothrock N, Keefe F, Callahan L, Lai JS. Development of a PROMIS item bank to measure pain interference. Pain. 2010 Jul;150(1):173-182. doi: 10.1016/j.pain.2010.04.025. PMID 20554116
- [Result] Davis, F. D. (1989). Perceived usefulness, perceived ease of use, and user acceptance of information technology. MIS Quarterly, 13, 319-340.
- [Result] Venkatesh, V. (2000). Determinants of perceived ease of use: Integrating perceived behavioral control, computer anxiety and enjoyment into the technology acceptance model. Information Systems Research, 11, 342-365.
- [Result] Venkatesh, V., & Bala, H. (2008). Technology Acceptance Model 3 and a research agenda on interventions. Decision Sciences, 39(2), 273-315. https://doi.org/10.1111/j.1540-5915.2008.00192.x
- [Derived] Remillard ET, Mitzner TL, Mumma KT. Tele Tai Chi for people aging with mobility disabilities: Novel methodology and structured adaptation approach. Contemp Clin Trials Commun. 2025 Aug 28;47:101543. doi: 10.1016/j.conctc.2025.101543. eCollection 2025 Oct. PMID 40969304